CLINICAL TRIAL: NCT06661980
Title: Effect of Dexmedetomidine on Brain Injury Patients
Brief Title: Dexmedetomidine on Brain Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DXM in brain Injury
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: All enrolled 60 patients will be mentioned as two groups; Group 1(n=30): are the patients who will receive dexmedetomidine. Group 2 (n=30): are the patients who represent the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Group (Active Comparator): 30 brain injury patients will treated with Dexmedetomidine 200 mcg/ 2 mL (Intravenous infusion).
  Interventions: Drug: Dexmedetomidine Injectable Solution
- Placebo Group (Placebo Comparator): 30 brain injury patients will treated with Placebo Normal Saline 2ml (Intravenous infusion).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine Injectable Solution — Dexmedetomidine 200 mcg/ 2 mL IV.
  Other Names: Dexmedetomidine
  Arms: Dexmedetomidine Group
Other: Placebo — Normal Saline 2ml IV.
  Other Names: NS
  Arms: Placebo Group

SUMMARY:
The aim of the study is to check whether dexmedetomidine has neuroprotective properties in brain injury patients. The enrolled 60 patients will be divided into two groups; Group 1(n=30): are the patients who will receive dexmedetomidine. Group 2 (n=30): are the patients who represent the control group.

DETAILED DESCRIPTION:
1. Approval will be obtained from the Research Ethics Committee of Faculty of Pharmacy, Damanhour University.
2. All participants must agree to take part in this clinical study and provide informed consent.
3. The required sample size will be calculated.
4. 60 Patients with brain injury will be enrolled from the intensive care department, Damanhour medical national institute.
5. Serum samples will be collected for measuring the biomarkers.
6. All enrolled 60 patients will be mentioned as two groups; Group 1(n=30): are the patients who will receive dexmedetomidine. Group 2 (n=30): are the patients who represent the control group.
7. All patients will be followed up during their stay in the intensive care department.
8. During their stay in the intensive care department, step 5 will be repeated.
9. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
10. Measuring outcomes: the primary outcome is measuring the neuroprotection provided by dexmedetomidine reflected by change in patients' symptoms, while secondary outcome is the change in the level of biomarkers from baseline to post-treatment.
11. Results, discussion, conclusion, and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* 60 Patients with brain injury with age ranging from 18 to 70 years, there are no limits to gender.

Exclusion Criteria:

* Patients with significant liver impairment
* Patients with known heart failure
* Patients with hypotension
* Patients with bradycardia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Glasgow Coma Scale (number) | 1 week
  GCS The highest possible 15, and the lowest is 3. A score of 15 means fully awake, responsive and have no problems with thinking ability or memory. Generally, having a score of 8 or fewer means a coma. The lower the score, the deeper the coma is.
length of intensive care department stay (days) | 1 month
  length of intensive care department stay.

SECONDARY OUTCOMES:
Neuron Specific Enolase (ng/ml) | 1 Week
  Biomarker (NSE)
tau protein (ng/L) | 1 Week
  Biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M. Mostafa, Prof., Study Chair — Tanta University
Locations (1):
- Damanhour Teaching Hospital, General Organization for Teaching Hospitals and Institutes., Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu Y, Zhou H, Zhang H, Sui Y, Zhang Z, Zou Y, Li K, Zhao Y, Xie J, Zhang L. The neuroprotective effect of dexmedetomidine and its mechanism. Front Pharmacol. 2022 Sep 20;13:965661. doi: 10.3389/fphar.2022.965661. eCollection 2022. PMID 36204225
- [Background] Isgro MA, Bottoni P, Scatena R. Neuron-Specific Enolase as a Biomarker: Biochemical and Clinical Aspects. Adv Exp Med Biol. 2015;867:125-43. doi: 10.1007/978-94-017-7215-0_9. PMID 26530364